CLINICAL TRIAL: NCT00982878
Title: The Penetration of Maraviroc Into the Central Nervous System in HIV-1 Infected Subjects on Stable Antiretroviral Therapy; a Phase I Pharmacokinetic Study
Brief Title: The Maraviroc Central Nervous System (CNS) Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Alan Winston, Reader and Honorary HIV consultant, Imperial College London
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-008437-10
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Results first posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: HIV Infections
Keywords: treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Maraviroc (Experimental)
  Interventions: Drug: Maraviroc

INTERVENTIONS:
Drug: Maraviroc — 150mg twice daily

SUMMARY:
The purpose of this study is to describe the Central Nervous System exposure of maraviroc in HIV-1 infected subjects receiving a stable antiretroviral regimen, including maraviroc, at steady state.

DETAILED DESCRIPTION:
15 HIV-1 infected subjects currently receiving stable antiretroviral therapy will be recruited. At study entry, within 14 days of screening procedures, subjects will commence maraviroc dosed at 150 mg twice daily. For the rest of study period antiretroviral therapy will comprise:

* Truvada™ one tablet once daily at 0900
* Kaletra™ two tablets twice daily 0900 and 2100
* maraviroc 150 mg twice daily at 0900 and 2100

Subjects will attend for regular clinic visits during study treatment phase.

On day 15, subjects will attend the unit in the morning prior to usual dosing time. Blood with be drawn to assess plasma maraviroc concentration pre dose and pre lumbar puncture. A lumbar puncture will be performed under standard aseptic techniques to asses CSF maraviroc concentration and routine CSF parameters.

On completion of this study visit, subjects will cease maraviroc, continue on their usual antiretroviral regimen and attend for a follow up visit 10 days later.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected males or females
* signed informed consent
* plasma HIV RNA < 50 copies/mL at screening and on at least one other occasion over the last 3 months
* currently receiving a stable antiretroviral regimen comprising of:

  * tenofovir 245 mg daily
  * emtricitabine 200 mg daily
  * a boosted protease inhibitor
* no previous protease inhibitor resistance documented on HIV-1 genotypic resistance testing
* Between 18 to 65 years of age, inclusive
* subjects in good health upon medical history, physical exam, and laboratory testing
* Female subjects who are heterosexually active and of childbearing potential (i.e., not surgically sterile or at least two years post menopausal) must practice contraception as follows from screening through completion of the study including 30 days following last dose of study drug:

  * barrier contraceptives (condom, diaphragm with spermicide)
  * IUD PLUS a barrier contraceptive
* Female subjects of childbearing potential must have a negative pregnancy test.
* Male subjects who are heterosexually active must use two forms of barrier contraception (e.g., condom with spermicide) during heterosexual intercourse, from screening through completion of the study including 30 days following last dose of study drug.
* Have no serologic evidence of active HBV infection evidenced by negative hepatitis B surface antigen and no serologic evidence of hepatitis C virus infection by a HCV antibody or HCV PCR.
* Have screening laboratory results (haematology, chemistry, and urinalysis) that fall within the normal range of the central laboratory's reference ranges unless the results have been determined by the Investigator to have no clinical significance

Exclusion Criteria:

* current alcohol abuse or drug dependence
* active opportunistic infection or significant co-morbidities including dementia
* current prohibited concomitant medication (as listed in section 4.1.4)
* Have a body mass index (BMI) > 32
* Contraindication to lumbar puncture examination. Such as:

  * Existing neurological diseases
  * Bleeding disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2010-07 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Winston, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Garvey L, Nelson M, Latch N, Erlwein OW, Allsop JM, Mitchell A, Kaye S, Watson V, Back D, Taylor-Robinson SD, Winston A. CNS effects of a CCR5 inhibitor in HIV-infected subjects: a pharmacokinetic and cerebral metabolite study. J Antimicrob Chemother. 2012 Jan;67(1):206-12. doi: 10.1093/jac/dkr427. Epub 2011 Oct 10. PMID 21987241

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Maraviroc
Started | 13
Completed | 12
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Maraviroc
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 4
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 12
Years since HIV diagnosis [Mean (Standard Deviation); unit: years] | 11 (4.6)
Baseline CD4 cell count [Mean (Standard Deviation); unit: cells/ul] | 503 (199)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28 (3.5)

OUTCOME MEASURES:

1. Primary Outcome: CSF (Cerebrospinal Fluid) : Plasma Ratio of Maraviroc 1H Magnetic Resonance Spectroscopy (1H-MRS)
Description: To describe the CNS exposure of maraviroc in HIV-1 infected subjects receiving a stable antiretroviral regimen, including maraviroc, at steady state.
  It were assessed by in vivo cerebral (1)H magnetic resonance spectroscopy ((1)H-MRS).
  Cerebral MRS imaging (T1- and T2-weighted images) was performed on a Phillips Achieva™ 1.5 Tesla magnetic resonance (MR) scanner (Phillips NV, Best, Netherlands) and studied by an experienced neuroradiologist
Time Frame: 15 days
Measure: Mean (Full Range); unit: ratio
Arm/Group | Maraviroc
Number analyzed (Participants) | 12
ratio | 1.01 [0.57 to 1.61]

2. Secondary Outcome: Number of Participants With Adverse Events
Description: To evaluate the short term safety and tolerability of maraviroc in HIV-1 infected subjects on stable antiretroviral therapy
Time Frame: 15 days
Measure: Count of Participants; unit: Participants
Arm/Group | Maraviroc
Number analyzed (Participants) | 12
Participants | 0

ADVERSE EVENTS:
Time Frame: 15 days
Arm/Group | Maraviroc
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes